CLINICAL TRIAL: NCT02692976
Title: A Randomized Phase IIa Study: Natural Dendritic Cells for Immunotherapy of Chemo-naive Metastatic Castration-resistant Prostate Cancer Patients
Brief Title: Natural Dendritic Cells for Immunotherapy of Chemo-naive Metastatic Castration-resistant Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2012-002531-29
Record Dates: First submitted 2015-09-30; First posted 2016-02-26 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2018-11

CONDITIONS: Prostatic Neoplasms; Immunotherapy; Dendritic Cells; Vaccines
Keywords: Castration-resistant prostate cancer; Dendritic Cells; Immunotherapy; Vaccines
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Myeloid dendritic cells (mDC) vaccinations (Experimental): Patients will be vaccinated intranodally three times biweekly with mDC (5x 106 cells; n=7, arm A). DC will be loaded with major histocompatibility complex (MHC) class I binding peptides of tumor antigens and NY-ESO-1 and MUC1 PepTivator® which covers the complete antigen. DC will be stimulated with protamine/mRNA and loaded with keyhole limpet hemocyanin (KLH) as an immune control.
  Interventions: Biological: mDC vaccination
- Plasmacytoid dendritic cells (pDC) vaccinations (Experimental): Patients will be vaccinated intranodally three times biweekly with pDC (3x 106 cells; n=7, arm B). DC will be loaded with MHC class I binding peptides of tumor antigens and NY-ESO-1 and MUC1 PepTivator® which covers the complete antigen. DC will be stimulated with protamine/mRNA.
  Interventions: Biological: pDC vaccination
- mDC and pDC vaccinations (Experimental): Patients will be vaccinated intranodally three times biweekly with the combination of mDC and pDC (5x 106 mDC/ 3x 106 pDC; n=7, arm C). DC will be loaded with MHC class I binding peptides of tumor antigens and NY-ESO-1 and MUC1 PepTivator® which covers the complete antigen. DC will be stimulated with protamine/mRNA and loaded with KLH (mDC only) as an immune control.
  Interventions: Biological: mDC and pDC vaccination

INTERVENTIONS:
Biological: mDC vaccination — Intranodal mDC vaccination
  Arms: Myeloid dendritic cells (mDC) vaccinations
Biological: pDC vaccination — Intranodal pDC vaccination
  Arms: Plasmacytoid dendritic cells (pDC) vaccinations
Biological: mDC and pDC vaccination — Intranodal mDC/pDC vaccination
  Arms: mDC and pDC vaccinations

SUMMARY:
Prostate cancer is the only type of cancer in which conventional dendritic cells (DC) treatment has a beneficial effect on the overall survival. In this study investigators aim to show immunologic efficacy of tumor-peptide loaded natural DC in metastatic castration-resistant prostate cancer patients (mCRPC).

The immunomonitoring will include:

1. functional response and tetramer analysis of delayed-type hypersensitivity infiltrating lymphocytes against tumor peptides and
2. type I interferon (IFN) gene expression in peripheral blood mononuclear cells, and
3. proliferative, effector cytokine- and humoral responses to keyhole limpet hemocyanin, a immunogenic protein providing T cell help.

The secondary objectives are the safety and feasibility of natural DC vaccinations, the influence on the quality of life during treatment with natural DC, and the clinical efficacy of treatment.

DETAILED DESCRIPTION:
Immunotherapy with DC vaccines Prevention of infectious diseases through immunization is one of the greatest achievements of modern medicine. Nonetheless, considerable challenges remain for improving the efficacy of existing vaccines for therapeutic immunizations for diseases such as cancer. More than 10 years ago the first groups introduced tumor antigen-loaded DC-based vaccines in the clinic. Effective immune responses and favorable clinical outcomes have indeed been observed. Thus far, mainly conventional in vitro generated monocyte-derived DCs (moDC) have been used in clinical trials worldwide. Long lasting tumor specific T cell-mediated immunological responses are clearly linked to increased progression free survival as well as overall survival.

However, moDC may not be the optimal source of DCs for DC vaccination studies, due to extensive culture periods and compounds required to obtain mature moDC. Two principal subsets of human blood DC, called plasmacytoid DC (pDC) and myeloid DC (mDC), are possibly a better alternative since they do not require extensive culture periods and are directly isolable from the peripheral-blood. Based on promising immunological and clinical outcome with pDC and mDC vaccinations in metastatic melanoma patients, further testing of these blood DC subsets is warranted. Based on these observations investigators are convinced that pDC and mDC employ different, and probably more optimal mechanisms to combat cancer. In addition, based on in vitro data and preclinical studies that suggest that natural DC act synergistically, investigators hypothesize that the combination of pDC and mDC may induce stronger anti-tumor immune responses as compared to pDC or mDC alone.

Immunotherapy in prostate cancer Prostate cancer is the most common noncutaneous cancer in men. In recent years novel therapies have been studied extensively. Prostate cancer is usually diagnosed in men above 65 years of age. Depending on the severity of the disease, current treatment options for prostate cancer consist of active surveillance, prostatectomy, radiation therapy, hormonal therapy, or chemotherapy. Up to one-third of patients with a localized tumor eventually fails on local therapy and progress to advanced-stage or metastatic disease within 10 years. Although the majority of patients initially respond to anti-androgens, most tumors become resistant within 14 to 30 months. For men with mCRPC the median survival in phase III studies range from 15 to 19 months. The chemotherapeutic drug docetaxel was for several years the only treatment option for mCRPC, resulting in a median overall survival benefit of two to three months compared to mitoxantrone. In the past five years second-line chemotherapy (cabazitaxel), second-generation androgen deprivation therapy (abiraterone acetate plus prednisone and enzalutamide), cellular immunotherapy (sipuleucel-T), and a targeted alpha emitter (radium-223 treatment) have expanded the treatment repertoire for mCRPC.

Sipuleucel-T, a DC-based vaccine for patients suffering from prostate cancer, has shown to be clinically effective and is approved by the Food and Drug Administration and European Medicines Agency for mCRPC patients. A major advantage of cellular immunotherapy when compared to chemotherapy, and even androgen deprivation therapy, is its low toxicity. Several other immunotherapeutic approached have been investigated and potential tumor antigens have been identified. Prostvac (vaccinia-prostate-specific antigen) was administered in a randomized phase II study with encouraging results. Ipilimumab had promising results in several phase II studies and in combination with a vaccine, such as GVAX. However, in a phase III study post-chemotherapy trial ipilimumab seemed not superior to placebo. Hence, only sipuleucel-T had clinical significant results in clinical trials.

The promising immunological and clinical outcome with pDC and mDC in metastatic melanoma warrants further testing of these blood DC in prostate cancer. In this study investigators aim to show proof-of-principle of natural DC immunogenicity in prostate cancer patients: induction/enhancement of tumor-specific T cells by mDC and induction of an IFN signature by pDC. Investigators will also get insight if combining subsets improves immunogenicity and clinical outcome. Hence, there is an urgent need for a potent treatment modality together with a solid predictive and prognostic biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years of age and older with confirmed (histologically or cytologically) adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
* Human leukocyte antigen (HLA)-A2.1 positive
* Asymptomatic or minimally symptomatic metastatic castration-resistant prostate cancer (mCRPC)
* Metastatic castrate-resistant disease defined as one or more of the following criteria that occurred while the patient was on androgen deprivation therapy:

  * Prostate-specific antigen (PSA)-progression defined by Prostate Cancer Working Group 2 (PCWG2) criteria by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination
  * Progression of nodal metastases defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 criteria or progression on successive magnetic resonance imaging lymphangiographies (MRLs)
  * Bone disease progression defined by two or more new lesions on bone scan as described in PCWG2 criteria
* Maintenance of castrate circumstances:

  * Ongoing primary androgen deprivation therapy (Gonadotropin-Releasing hormone agonist or antagonist) or bilateral orchiectomy
  * Serum testosterone level ≤ 1.73 nmol/L (50 ng/dL) at screening visit
* PSA value ≥ 2 ng/ml
* Absence of visceral metastases, malignant ascites or pleural effusion
* Clinical absence of brain metastases
* Inclusion within three months after the moment of manifestation of progressive disease as defined above
* Chemotherapy naive
* Life expectancy ≥ 6 months
* World Health Organization/Eastern Cooperative Oncology Group performance status 0-1 (Karnofsky index 100-70)
* White blood cells >2.0x109/l, neutrophils >1.5x109/L, lymphocytes >0.8x109/L, platelets >100x109/L, hemoglobin >5,6 mmol/L (9.0 g/dL), serum creatinine <150 µmol/L, aspartate aminotransferase/alanine aminotransferase <3 x upper limit of normal (ULN), serum bilirubin <1.5 x ULN (exception: Gilbert's syndrome is permitted)
* Expected adequacy of follow-up
* Written informed consent

Acceptable concomitant therapy:

* The use of oral or intravenous bisphosphonates
* Radiotherapy for pain relief in patients with bone metastases may be used as a treatment modality, but the need for a radiotherapeutic intervention during the study will be documented as an skeletal-related event (SRE)
* Inhaled corticosteroids and topical creams for small body areas are permitted

Exclusion Criteria:

* Hypercalcemia
* History of any second malignancy in the previous five years, with the exception of adequately treated basal cell carcinoma
* Known allergy to shell fish
* Heart failure (New York Heart Association class III/IV)
* Serious active infections
* Active hepatitis B, C or HIV infection
* Active syphilis infection
* Autoimmune diseases (exception: vitiligo is permitted)
* Organ allografts
* An uncontrolled co-morbidity, e.g. psychiatric or social conditions interfering which participation
* Previous treatment with sipuleucel-T,PROSTVAC, GVAX, chemotherapy, ipilimumab or denosumab (previous treatment with abiraterone acetate, ketoconazole or enzalutamide is permitted)
* Treatment with flutamide, bicalutamide, or nilutamide within four weeks of study enrollment
* Prior radiotherapy within four weeks prior to planned vaccination or presence of treatment-related toxicity
* Continued use of non-steroidal anti-inflammatory drugs
* Concurrent use of systemic corticosteroids > 10 mg daily prednisone equivalent
* Requirement of opiate use for cancer-related pain (at screening)
* Any serious clinical condition that may interfere with the safe administration of DC vaccinations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-03-06 (Actual)

PRIMARY OUTCOMES:
The immunogenicity of tumor-peptide loaded natural blood dendritic cells (myeloid DC, plasmacytoid DC and the combination of mDC/pDC) in metastatic castration-resistant prostate cancer (mCRPC) patients | 18 months
  a.functional response and tetramer analysis of delayed-type hypersensitivity infiltrating lymphocytes against tumor peptides.
The immunogenicity of tumor-peptide loaded natural blood dendritic cells (myeloid DC, plasmacytoid DC and the combination of mDC/pDC) in metastatic castration-resistant prostate cancer (mCRPC) patients | 18 months
  b.type I interferon (IFN) gene expression in peripheral blood mononuclear cells.
The immunogenicity of tumor-peptide loaded natural blood dendritic cells (myeloid DC, plasmacytoid DC and the combination of mDC/pDC) in metastatic castration-resistant prostate cancer (mCRPC) patients | 18 months
  c.proliferative, effector cytokine- and humoral responses to keyhole limpet hemocyanin, a immunogenic protein providing T cell help.

SECONDARY OUTCOMES:
Treatment-related adverse events assessment by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | 18 months
  Number of participants with treatment-related adverse events as assessed by CTCAE version 4.0 and establishing the feasibility of the st-udy protocol by looking at the enrollment duration. The CTCAE version 4.0 displays Grades 1 through 5 with unique clinical descriptions of severity for each adverse event (AE) based on this general guideline:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Quality of life measurement by EORTC-QLQ-C30 | 18 months
  Quality of life measured with EORTC-QLQ-C30 questionnaire. A higher functional scale score represents a higher level of functioning. A high score for Global Health Status represents a high HRQoL. A high symptom or single-item score represents a high symptomatology level. A clinically relevant difference was defined by a mean change of at least 10 points on a scale score
Quality of life measurement by EORTC-QLQ-PR25 | 18 months
  Quality of life measured with EORTC-QLQ-PR25 questionnaire. A higher score on functioning-related domains is indicative for better functioning, where a higher symptom-related domain score is indicative for more symptomatology. Sexual functioning questions required reversing of the response categories for 3 of 4 questions (question number 23-25). In line with the EORTC-QLQ-C30, a clinically relevant difference was defined by a mean change of at least 10 points on a scale scores.
Quality of life measurement by BDI (PC) | 18 months
  Quality of life measured with BDI (PC) questionnaire. The BDI-PC questionnaire is one of the rating scales for identifying a mood disorder in medical outpatients. BDI-PC is a seven item questionnaire with scores ranging from 0 to 21. Scores of 4 or higher are suggestive for a clinical relevant depression.
Quality of life measurement by CIS20-R | 18 months
  Quality of life measured with CIS20-R questionnaire. The CIS-20R is a self-report questionnaire assessing 20 items incarcerating four fatigue dimensions (subjective experience of fatigue (CIS1), reduction in concentration (CIS2), reduction in motivation (CIS3) and reduction in activity (CIS4)). Patients rated the extent to which each statement was true for the previous two weeks on a 7-category scale (ranging from score 1 'Yes, that is true' to 7 'No, that is not true'). A CIS1 score of 35 of higher indicates severe fatigue. A score between 27 and 35 represents an increased risk for fatigue.
Prostate-specific antigen (PSA)-progression | every 6 weeks, up to 24 months
  PSA progression will be defined according to the Prostate Cancer Clinical Trials Working Group 2 (PCWG2) criteria.
Progression Free Survival (PFS) | every 6 weeks, up to 24 months
  To evaluate PFS: serum PSA value will be determined every 6 weeks and a magnetic resonance imaging lymphangiography (MRL) will be performed every 3 months (combined with a 68Ga-PSMA-PET/CT scan at t=0 and t=3 months, and for long responders to therapy at t=12 months and t=24 months). PFS is defined as the time from randomization to the detection of progressive disease on MRL/68-Ga-PSMA-PET/CT scan or immune-related progressive disease, including new measurable lesions reported on successive MRLs. According to the PCWG2 criteria. In case of disease progression during vaccination the patient will be withdrawn from the study. In case of stable disease after three rounds of vaccinations follow-up with MRL will be performed until 24 months after study enrollment.
Overall Survival (OS) | 2 years
  OS will be determined at the end of study follow-up. The patient's general practitioner will be contacted for OS analysis.
Time to opiate use | every 3 months, up to 24 months
Time to skeletal-related event (SRE) | every 3 months, up to 24 months
  Defined by MRI
World Health Organization (WHO) performance score decline | every 6 weeks, up to 24 months
  Defined by 1 or more point decline in WHO/ECOG performance score
Time to chemotherapy initiation after mDC/pDC vaccinations | every 6 weeks, up to 24 months
Radiologic profression-free survival | MRI: every 3 months; 68-Ga-PSMA-PET/CT scan: t=0, 3, 12 en 24 months, up to 24 months.
  Determined on MRI scans/68-Ga-PSMA-PET/CT scan
Feasibility of the natural DC vaccination trial | 18 months
  Feasibility of participant recruitment and the collection of immunological and clinical data within the time frame of 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Winald R Gerritsen, MD PhD, Principal Investigator — Radboudumc, dep of Medical Oncology; Fred Witjes, MD PhD, Principal Investigator — Radboudumc, dep of Urology; Jolanda IM de Vries, PhD, Study Director — Radboudumc, dep of Tumor Immunology, laboratory study coordinator
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after all clinical and immunological data collection and analysis in a scientific publication.

REFERENCES:
- [Derived] Westdorp H, Creemers JHA, van Oort IM, Mehra N, Hins-de Bree SM, Figdor CG, Witjes JA, Schreibelt G, de Vries IJM, Gerritsen WR, Ottevanger PB. High Health-Related Quality of Life During Dendritic Cell Vaccination Therapy in Patients With Castration-Resistant Prostate Cancer. Front Oncol. 2020 Oct 26;10:536700. doi: 10.3389/fonc.2020.536700. eCollection 2020. PMID 33194595
- [Derived] Westdorp H, Creemers JHA, van Oort IM, Schreibelt G, Gorris MAJ, Mehra N, Simons M, de Goede AL, van Rossum MM, Croockewit AJ, Figdor CG, Witjes JA, Aarntzen EHJG, Mus RDM, Bruning M, Petry K, Gotthardt M, Barentsz JO, de Vries IJM, Gerritsen WR. Blood-derived dendritic cell vaccinations induce immune responses that correlate with clinical outcome in patients with chemo-naive castration-resistant prostate cancer. J Immunother Cancer. 2019 Nov 14;7(1):302. doi: 10.1186/s40425-019-0787-6. PMID 31727154